CLINICAL TRIAL: NCT03523598
Title: Potassium Nitrate Influence on Post in Office Bleaching Sensitivity: a Triple Blinded Randomized Clinical Trial
Brief Title: Potassium Nitrate and Post-bleaching Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sergipe (Other)
Collaborators: Johnny Alexandre Oliveira Tavares (Unknown)
Responsible Party: Principal Investigator, Flavia Pardo Salata Nahsan, Clinical Professor, Universidade Federal de Sergipe
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFSergipe.
Record Dates: First submitted 2018-04-09; First posted 2018-05-14 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Medicaments Substances in Therapeutic Use

STUDY DESIGN:
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo gel + Normal Toothpaste (Placebo Comparator): The patient will receive the application of placebo gel on vestibular surface teeth, for 10 minutes and will use the normal toothpaste (Colgate).
  Interventions: Other: Placebo gel + Normal Toothpaste
- Placebo Gel + Potassium Nitrate Toothpaste (Experimental): The patient will receive the application of placebo gel on vestibular surface teeth, for 10 minutes and will use the Potassium nitrate toothpaste (Sensodyne).
  Interventions: Other: Placebo Gel + Potassium Nitrate Toothpaste
- Potassium Nitrate Gel + Normal Toothpaste (Experimental): The patient will receive the application of 5% Potassium nitrategel on vestibular surface teeth, for 10 minutes and will use the normal toothpaste (Colgate).
  Interventions: Other: Potassium Nitrate Gel + Normal Toothpaste

INTERVENTIONS:
Other: Placebo gel + Normal Toothpaste — * 15 days before and during the period of bleaching sessions: Tooth paste used will be normal (Colgate).
  * Teeth will be cleaned using rubber cups associated to pumice and water;
  * Relative isolation with roller cotton will be done;
  * Prior to each bleaching session, the patients will receive the placebo gel application on vestibular surface, for 10 minutes.
  * Gingival dam will be performed using a fluid resin.
  * A 35% hydrogen peroxide based bleaching agent will applied on the vestibular surface of teeth, remaining for 40 minutes.
  Arms: Placebo gel + Normal Toothpaste
Other: Placebo Gel + Potassium Nitrate Toothpaste — * 15 days before and during the period of bleaching sessions: Tooth paste used will be normal tooth paste (Colgate).
  * Teeth will be cleaned using rubber cups associated to pumice and water;
  * Relative isolation with roller cotton will be done;
  * Prior to each bleaching session, the patients will receive the 5% Potassium Nitrate gel application on vestibular surface, for 10 minutes.
  * Gingival dam will be performed using a fluid resin.
  * A 35% hydrogen peroxide based bleaching agent will applied on the vestibular surface of teeth, remaining for 40 minutes.
  Arms: Placebo Gel + Potassium Nitrate Toothpaste
Other: Potassium Nitrate Gel + Normal Toothpaste — * 15 days before and during the period of bleaching sessions: Tooth paste used will be Potassium Nitrate containing (Sensodyne).
  * Teeth will be cleaned using rubber cups associated to pumice and water;
  * Relative isolation with roller cotton will be done;
  * Prior to each bleaching session, the patients will receive the placebo gel application on vestibular surface, for 10 minutes.
  * Gingival dam will be performed using a fluid resin.
  * A 35% hydrogen peroxide based bleaching agent will applied on the vestibular surface of teeth, remaining for 40 minutes.
  Arms: Potassium Nitrate Gel + Normal Toothpaste

SUMMARY:
This study will determine the effectiveness of the use of desensitivity gels prior in office bleaching on risk and intensity of tooth sensitivity caused by in-office bleaching using 35% hydrogen peroxide and using different types of potassium nitrate. Materials and Methods: Seventy five patients will be selected for this triple-blind, randomized, cross-over, placebo-controlled clinical trial. 10 minutes prior to bleaching procedure, patients will receive the the potassium nitrate 2% or placebo gel application on vestibular surface and Toothpaste 15 days before start the bleaching procedure (group 1: placebo gel + Colgate toothpaste; Group 2: Placebo gel + Nitrate toothpaste Sensodyne and Group 3: Potassium Nitrate + Colgate toothpaste). The whitening treatment with 35% hydrogen peroxide will be carried out in two sessions with a 7-day interval.

Tooth sensitivity will be assessed before, during and 24 hours after the procedure using analog visual and verbal scales. Color alteration will be assessed by a Vita Guide scale at the end of the last session. Relative risk to sensitivity will be calculated and adjusted by session; while comparison of overall risk will performed by McNemar's test. Data on the sensitivity level and color shade will be subjected to the Friedman, Wilcoxon (α = 0.05). If necessary, multiple comparation will be done using Tukey's test.

DETAILED DESCRIPTION:
This study will be a randomized, triple-blinded, placebo-controlled clinical trial, and split mouth study design.

The patients included will be submitted to two in-office bleaching sessions receiving the potassium nitrate 5% or placebo gel (prior the bleaching session, for 10 minutes), associated to normal toothpaste or potassium nitrate containing toothpaste (15 days prior and during the bleaching procedure).

A delay of 1 week between the sessions will be established.

Participants:

Patients included in this clinical trial will be between 18 and 29 years old with good oral health, all anterior tooth healthy and to agree with TCLE (Term of Free and Informed Consent). Only patients presenting all six upper anterior teeth with shade mismatching with 2.5 M2 (VitaClassicalscale, Vita-Zahnfabrik, Bad Sackingen, Germany).

Patients with any of the six upper anterior teeth with caries, restoration, severe discoloration (e.g., stains caused by tetracycline), enamel hypoplasia, gingival recession, dentin exposure, pulpitis, or endodontics will be excluded. Participants submitted to previous bleaching procedures, presenting prior tooth sensitivity, known allergy to any component of medication used in the study, pregnant or breastfeeding, lack the tretament will be also excluded.

Sample Size Calculation:

The sample calculation will be based on the primary binary outcome (sensitivity risk 24 hours after the procedure) for superiority trial. Power of the test will be set at 80%, considering a type I error of 0.05; risk to tooth sensitivity for control and experimental group of 25,2% with reduction of 60%. The calculation resulted in 75 patients.

Randomization:

A randomized list will be computer-generated by a person not involved in intervention or evaluation. The participants were defined as blocks in the randomization process, where the sequence of treatment (placebo or etodolac) will be randomly set for each block by using computer-generated tables (www.sealedenvelope.com). The sequence will be inserted into sealed envelopes numbered from 1 to 75 that were opened by the operator only at the moment of the intervention. The patients were numbered according to the sequence of enrollment. Neither the participant nor the operator will know the group allocation determining blinding to the protocol.

Baseline evaluation:

Prior to bleaching procedure, the teeth will be cleaned using rubber cups associated to pumice and water. The shades of six upper anterior teeth will be assessed on a baseline using the Vita classical guide scale.

Intervention:

Prior to each bleaching session, the patients will receive the potassium nitrate 2% or placebo Gel for 10 minutes. Also, Normal and potassium nitrate toothpaste will be used before and during the bleaching tretament, as follows: group 1: placebo gel + Colgate toothpaste; Group 2: Placebo gel + Nitrate toothpaste Sensodyne and Group 3: Potassium Nitrate + Colgate toothpaste.

Neither the operators responsible for intervention and evaluation nor the patients knew the content which treatment will be done.

A light-cured resin dam will be applied on the gingival tissue corresponding to the teeth to be bleached.

A 35% hydrogen peroxide based bleaching agent (DFL) will be mixed and applied on the vestibular surface of teeth, remaining for 40 minutes. After this time, the bleaching agent will be removed. A second session will be carried out after 1 week following the same procedures.

Evaluations:

The tooth sensitivity reported by patients will be assessed using a visual analog scale (VAS) and verbal rating scale (VRS). The VAS consisted of a scale 10 cm in length ranging from green (absence of pain) to red (unsupportable pain). The patient set his or her level of sensitivity by pointing to the color corresponding to this level, while the distance from this point to the green border will be recorded. For VRS, the patient reported his or her level of sensitivity based on scores: 0 = none, 1 = light, 2 = moderate, 3 = considerable and 4 = severe. The tooth sensitivity will be assessed during the bleaching, immediately after bleaching agent removal and after 24 hours. For this last assessment, only the VRS will be used. Tooth sensitivity will be measure: baseline, at 40 minutes during the bleaching procedure, after the bleaching procedure and 24 hours after. One week after each session the tooth color will be evaluated again using the same procedure described previously.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this clinical trial will be between 18 and 29 years old with good oral health;
* All anterior tooth healthy
* To agree with TCLE (Term of Free and Informed Consent).
* Only patients presenting all six upper anterior teeth with shade mismatching with 2.5 M2 (VitaClassicalscale, Vita-Zahnfabrik, Bad Sackingen, Germany).

Exclusion Criteria:

* Patients with any of the six upper anterior teeth with caries
* Restoration in anterior tooth, severe discoloration (e.g., stains caused by tetracycline), enamel hypoplasia, gingival recession, dentin exposure, pulpitis, or endodontics will be excluded.
* Participants submitted to previous bleaching procedures
* Presenting prior tooth sensitivity
* known allergy to any component of medication used in the study
* being pregnant or breastfeeding.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2018-05-26 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Risk to the tooth sensitivity (VAS) | During the bleaching treatment
  The tooth sensitivity will be assessed using a Visual analogue (VAS) scale. VAS consisted of a 10-cm scale 0 (no sensitivity) 10 (unbearable sensitivity). A slightly air-stream will be applied over the buccal surfaces of the central incisors, and the patients will record their sensitivity perception by pointing with a pen on the scale. The distance between the marking and the border of scale, relative to the absence of sensitivity will be measured. The measurements will be scored according to the distance from 0, using a digital caliper. The risk of tooth sensitivity will be determined by relative risk assessed by ratio between absolute risk of experimental condition by those observed in control. The 95% confidence interval will be calculated.
Risk to the tooth sensitivity (VRS) | During the bleaching treatment
  The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe. Score different from 0 will determine presence of sensitivity.The risk of tooth sensitivity will be determined by relative risk assessed by ratio between absolute risk of experimental condition by those observed in control. The 95% confidence interval will be calculated.

SECONDARY OUTCOMES:
Level of tooth sensitivity (VAS) | During the bleaching treatment
  The tooth sensitivity will be assessed using a Visual analogue (VAS) scale. VAS consisted of a 10-cm scale 0 (no sensitivity) 10 (unbearable sensitivity). A slightly air-stream will be applied over the buccal surfaces of the central incisors, and the patients will record their sensitivity perception by pointing with a pen on the scale. The distance between the marking and the border of scale, relative to the absence of sensitivity will be measured. The measurements will be scored according to the distance from 0, using a digital caliper. The risk of tooth sensitivity will be determined by relative risk assessed by ratio between absolute risk of experimental condition by those observed in control. The 95% confidence interval will be calculated.
Level of tooth sensitivity (VRS) | During the bleaching treatment
  The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe. Score different from 0 will determine presence of sensitivity.The risk of tooth sensitivity will be determined by relative risk assessed by ratio between absolute risk of experimental condition by those observed in control. The 95% confidence interval will be calculated.
Risk after tooth sensitivity- after the procedure (VAS) | 24 hours after the Bleaching procedure
  The tooth sensitivity will be assessed using a Visual analogue (VAS) scale. VAS consisted of a 10-cm scale 0 (no sensitivity) 10 (unbearable sensitivity). A slightly air-stream will be applied over the buccal surfaces of the central incisors, and the patients will record their sensitivity perception by pointing with a pen on the scale. The distance between the marking and the border of scale, relative to the absence of sensitivity will be measured. The measurements will be scored according to the distance from 0, using a digital caliper. The risk of tooth sensitivity will be determined by relative risk assessed by ratio between absolute risk of experimental condition by those observed in control. The 95% confidence interval will be calculated.
Risk after tooth sensitivity- after the procedure (VRS) | 24 hours after the Bleaching procedure
  The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe. Score different from 0 will determine presence of sensitivity.The risk of tooth sensitivity will be determined by relative risk assessed by ratio between absolute risk of experimental condition by those observed in control. The 95% confidence interval will be calculated.
Level of tooth sensitivity - after the procedure (VAS) | 24 hours after the Bleaching procedure
  The tooth sensitivity will be assessed using a Visual analogue (VAS) scale. VAS consisted of a 10-cm scale 0 (no sensitivity) 10 (unbearable sensitivity). A slightly air-stream will be applied over the buccal surfaces of the central incisors, and the patients will record their sensitivity perception by pointing with a pen on the scale. The distance between the marking and the border of scale, relative to the absence of sensitivity will be measured. The measurements will be scored according to the distance from 0, using a digital caliper. The risk of tooth sensitivity will be determined by relative risk assessed by ratio between absolute risk of experimental condition by those observed in control. The 95% confidence interval will be calculated.
Level of tooth sensitivity - after the procedure (VRS) | 24 hours after the Bleaching procedure
  The tooth sensitivity will be evaluated using a 5-point Verbal rating scale (VRS), where 0 = none, 1 = mild, 2 = moderate, 3 = considerable and 4 = severe. Score different from 0 will determine presence of sensitivity.The risk of tooth sensitivity will be determined by relative risk assessed by ratio between absolute risk of experimental condition by those observed in control. The 95% confidence interval will be calculated.
Bleaching Effectiveness | Before the bleaching procedures (baseline) and end of the treatment (an average of 14 days)
  The color evaluation will be performed classical Vita guide.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sergipe, Aracaju, Sergipe, Brazil

IPD SHARING:
Plan to Share IPD: No